CLINICAL TRIAL: NCT05736094
Title: Dual-frequency Ultrasound for Detection of Prostate Cancer
Brief Title: Ultrasound for Detection of Prostate Cancer
Acronym: SURF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); University of Oslo (Other); The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Wolfgang Lilleby, Principal Investigator, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 248446; 313778 (Other Grant/Funding Number: The Research Council of Norway)
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dual-frequency ultrasound (Other): Dual-frequency ultrasound for detection of prostate cancer
  Interventions: Device: SURF

INTERVENTIONS:
Device: SURF — Dual-frequency ultrasound

SUMMARY:
Clinical proof of concept of dual-frequency ultrasound imaging for detection and visualization of prostate cancer.

DETAILED DESCRIPTION:
Prospectively recruited patients before prostatectomy and/or definitive radiotherapy will be included in the study. Dual-frequency ultrasound imaging will be compared to standard transrectal ultrasound and MRI. Imaging of primary tumor with dual-frequency ultrasound technology including the use of microbubble contrast-media.

A prostate biopsy and blood sample will be taken from each patient, for histopathology and explorative biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years onwards
* Signed written informed consent to perform rectal and transperineal ultrasound

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only men will be included as prostate cancer does not appear in women
Enrollment: 11 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Clinical proof of concept of dual-frequency ultrasound imaging for detection and visualization of prostate cancer. | 1 day
  Sensitivity and specificity outcome measures
Clinical proof of concept of dual-frequency ultrasound imaging for detection and visualization of prostate cancer. | 1 day
  Comparing dual-frequency ultrasound, shear waves ultrasound, CEUS to MRI and histopathological findings

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Lilleby, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway